CLINICAL TRIAL: NCT03688737
Title: The Effect of Adjunctive Use of Low Level Laser (LLL) After Surgical Correction of Isolated Cleft Palate Versus Surgical Correction Without LLL in Healing Process
Brief Title: Low Level Laser in Isolated Cleft Palate Repair Versus Surgical Correction Without LLL in Healing Process
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, El noman Mohamed Kamal El shafie, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 172162009
Record Dates: First submitted 2018-09-24; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Cleft Palate Children; Laser
Keywords: low level laser , cleft palate , healing
MeSH Terms: conditions — Cleft Palate | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either control or study group in the ratio of 1:1 using random number table.
Who Masked: Participant
Masking Description: Single blinded study. Blinding to the patient will be ensured by masking the instruments during the follow up. The patient will be informed of the steps of the follow up (as mentioned in the consent form) without getting into details of the method of follow up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): A) Control group:
  Has Surgical procedures "von Langenbeck technique " to repair cleft palate and will come for follow up visit at day of surgery, 1st day and 3rd day for placebo device like LLL and come for follow up visits at 5th day ,2 weeks, month and 3 months postoperative
  Interventions: Other: placebo
- study group (Active Comparator): B) Study group:
  This group will be subjected to the same surgical procedure "von Langenbeck technique "to repair cleft palate but low level laser Therapy will be at day of surgery, 1st day and 3rd day and come for follow up visits at 5th day ,2 weeks, month and 3 months postoperative
  Interventions: Other: low level laser

INTERVENTIONS:
Other: low level laser — LLLT with wavelength (λ) of (600 nm to 700nm), The laser will be held 1 cm away from the surface of the target tissue, the irradiated area is 0,5 cm2.The area of impact is the surgical wound zone and the neighboring 0,5-1,0 cm of the adjacent oral mucosa for 1min and 22sec, at day of surgery, 1st day and 3rd day and come for follow up visits at 5th day ,2 weeks, month and 3 months postoperative
  Other Names: wavelength (λ) of (600 nm to 700nm)
  Arms: study group
Other: placebo — placebo like device as it like low level laser device shape but with no effect to blind the intervention
  Arms: control group

SUMMARY:
Does the use of low level laser (LLL) after surgical correction of cleft palate improve healing and decrease incidence of oronasal fistula?

DETAILED DESCRIPTION:
Primary objective:

To evaluate the effect of adjunctive use of LLL after surgical correction of cleft palate in improving healing among children with cleft palate Secondary objectives To evaluate the effect of adjunctive use of LLL after surgical correction of cleft palate in decreasing incidence of oronasal fistula after surgical repair among children with cleft palate Study group: Will use LLL after surgical correction of cleft palate at day of surgery, 1st day and 3rd day Control group: Surgical correction of cleft palate without Adjunctive use of LLL

Inclusion criteria:

1. Age: between 6 to 18 months of age
2. Patient has isolated cleft palate

Exclusion criteria:

1. Systemic disease
2. Hematological disorder Outcome: Outcome measure (s) (1ry, 2ry) 1ry: healing assessment 2ry: occurrence of oronasal fistula

ELIGIBILITY:
Inclusion Criteria:

1. Age: between 6 to 18 months of age
2. Patient has isolated cleft palate

Exclusion Criteria:

1. Systemic disease
2. Hematological disorder

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
wound healing | 2 years
  healing by days to closure

SECONDARY OUTCOMES:
occurrence of oronasal fistula | 3 months
  Postoperative complications; mainly oronasal fistula by; clinical observation: inspection, clinical signs: regurgitation of food or drink

IPD SHARING:
Plan to Share IPD: No